CLINICAL TRIAL: NCT00819637
Title: A Pilot Study to Determine the Most Effective Dose of Arformoterol for Treating Acute Asthmatic Patients Presenting to the Emergency Department and to Evaluate Its Side Effect and Safety Profile When Used in This Clinical Situation.
Brief Title: A Pilot Study to Determine the Most Effective Dose of Arformoterol for Treating Acute Asthmatic Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll r/t study design & staffing issues. The trial terminated.
Sponsor: Henry Ford Health System (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASRC947
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Results first posted 2010-06-29 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Acute Asthma
Keywords: Acute asthma; Arformoterol; Long acting beta agonists
MeSH Terms: interventions — Formoterol Fumarate; Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arformoterol 3 doses (Experimental)
  Interventions: Drug: arformoterol (RR formoterol)
- Arformoterol 1 dose, placebo 2 doses (Experimental)
  Interventions: Drug: arformoterol (RR formoterol); Drug: placebo
- Levalbuterol 3 doses (Active Comparator)
  Interventions: Drug: levalbuterol

INTERVENTIONS:
Drug: arformoterol (RR formoterol) — Group 1 will receive nebulized arformoterol 15 ug every 20 minutes for 3 doses.
  Group 2 will receive nebulized arformoterol 15 ug first dose and then placebo every 20 minutes for 2 doses.
  Other Names: Brovana
  Arms: Arformoterol 1 dose, placebo 2 doses; Arformoterol 3 doses
Drug: placebo — Group 2 will receive nebulized arformoterol 15 ug first dose and then placebo every 20 minutes for 2 doses.
  Arms: Arformoterol 1 dose, placebo 2 doses
Drug: levalbuterol — Group 3 will receive nebulized levalbuterol 1.25 mg every 20 minutes for 3 doses.
  Other Names: Xopenex
  Arms: Levalbuterol 3 doses

SUMMARY:
The purpose of this study is to determine the best dose of nebulized arformoterol, a quick onset but long acting beta agonist, for use in treating acute bronchospasm in asthmatics presenting to the the Emergency Department. Also this study will evaluate the side effect and safety profile of arformoterol when used in this situation.

DETAILED DESCRIPTION:
Acute bronchospasm associated with exacerbations of asthma is a common problem. Currently the mainstay of treatment is inhalation albuterol, either levalbuterol or racemic mixture, in repetitive fashion depending on the resolution of the airways obstruction. Formoterol is a long-acting (>12 hours) selective beta2-agonist that has a very rapid onset of bronchodilatation (<3 minutes and thus similar to that produced by albuterol). Patients with acute bronchospasm could benefit from the prn use of formoterol as they would receive acute relief of their symptoms and this would last for a prolonged time period. Additionally formoterol has been reported to be 28-109 times as potent as albuterol and safe at doses of 54ug in healthy subjects and asthmatics. Racemic formoterol structurally has 2 chiral centers and thus is composed of 4 enantiomers. The RR form (or arformoterol) is the active bronchodilator and it is not clear what the physiologic actions of the other 3 enantiomers are. This study is the first to evaluate nebulized arformoterol solution for therapy of acute asthmatics presenting to the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* FEV1 between 20 and 60% predicted after having received 5 mg of albuterol and 0.5 mg of atrovent as nebulized standard of care therapy
* Male or female between the ages of 18 and 45
* Asthma diagnosed by a physician and present for at least 6 months
* oxygen saturation greater or equal to 90% on room air
* Non smoker or < 10 pack-year history
* No other cause for wheezing/sob as determined by the treating physician

Exclusion Criteria:

* Clinical evidence or history of hepatic, renal, cardiovascular, GI, endocrine, metabolic or CNS disease which might interfere with the conduct of the study
* Acute respiratory failure or other significant pathology of the pulmonary system
* Female subjects who are pregnant or lactating
* Currently receiving therapy for a psychiatric disorder
* Subjects with a known sensitivity to formoterol (racemic or RR) or albuterol (racemic or lev)
* History of hospitalization for asthma within 2 months or treatment for acute asthma in an ED within 2 weeks of study entry
* Past or current use of disallowed medications
* Participation in an investigational study within 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Nowak, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital Emergency Department, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open for enrollment from 1/8/09 until 11/19/09. Location was Henry Ford Hospital Emergency Department
Period: Overall Study
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Started | 2 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was closed after 2 patients were enrolled but the study data was not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 2 |  |  | 2
  >=65 years | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: The Averaged Mean Percent Change From Baseline FEV1 and PEFR (Percent Predicted and Absolute) After the 3 Doses of Study Drug
Time Frame: 1 hour
Population: Study was terminated after two patients enrolled. Data not collected.
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Most Effective Dose of Inhalation Arformoterol for Treating Acute Bronchospasm in Asthmatics by Evaluating the Averaged Mean Percent Change From Baseline % Predicted FEV1 After 3 Doses of Study Medication in Each of the 3 Groups
Description: The study was terminated early and therefore secondary outcome measures were not obtained.
Time Frame: 1 hour
Population: The study was terminated early and therefore outcome measures were not obtained.
Groups:
- Arformoterol 1 Dose, Placebo 2 Doses; Arformoterol 3 Doses; Levalbuterol 3 Doses: Not Measured
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Treated With Arformoteral in Acute Asthma Exacerbation as a Measure of Safety and Tolerability.
Description: The study was terminated early and therefore secondary outcome measures were not obtained.
Time Frame: 5 hours
Population: The study was terminated early and therefore outcome measures were not obtained.
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: The Mean Percent Change From Baseline in the FEV1 and PEFR (Absolute and Percent Predicted) Following Each Dose of Study Drug
Time Frame: 1 hour
Population: The study was terminated early, therefore outcome measures were not obtained.
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: The Mean Change From Baseline in the FEV1 and PEFR (Absolute and Percent Predicted) Following Each Dose of Study Drug
Description: The study was terminated early and therefore secondary outcome measures were not obtained.
Time Frame: 1 hour
Population: The study was terminated early and therefore outcome measures were not obtained
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: The Peak Change (Liters) and Peak Percent Change From Baseline in the FEV1 and PEFR (Absolute and Percent Predicted) Following Each Dose of Study Drug
Time Frame: 1 hour
Population: The study was terminated early and therefore outcome measures were not obtained
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: The Time to Onset of a 15% Improvement in FEV1 for Each Dose (Individual and Cumulative) and Total Dose of Study Medication to Reach This
Time Frame: 5 hour
Population: The study was terminated early and therefore outcome measures were not obtained
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: The Time Required to Achieve a FEV1 and PEFR > 60% Predicted for Each Dose (Individual and Cumulative)
Time Frame: 5 hours
Population: The study was terminated early and therefore outcome measures were not obtained
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Percent of Responders (Defined as Those Discharged Following Treatment Who Did Not Require Additional Therapy in the ED)
Description: The 2 subjects enrolled were both discharged home after study protocol completion, with no further treatment required in the ED setting.
Time Frame: 5 hours
Population: The study was terminated early and therefore outcome measures were not obtained
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Percent of Patients in Each Group Requiring Additional Therapies After the First Hour of Study Drug Treatments
Description: 2 subjects were enrolled. Neither required additional asthma treatment after the 1st hour of study drug teatments.
Time Frame: 5 hours
Population: The study was terminated early and therefore outcome measures were not obtained.
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: All of the Primary and Secondary Endpoints Partitioned by the Presenting PFT in Quartiles and the Presenting S Albuterol Levels in Quartiles
Time Frame: 5 hours
Population: The study was terminated early and therefore outcome measures were not obtained
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Pharmacokinetics of Arformoterol in This Clinical Setting
Time Frame: 5 hours
Population: The study was terminated early and therefore outcome measures were not obtained.
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arformoterol 1 Dose, Placebo 2 Doses | Arformoterol 3 Doses | Levalbuterol 3 Doses
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes